CLINICAL TRIAL: NCT05236283
Title: Duration of Antimicrobial Treatment for Bloodstream Infections in Swiss Critically Ill Patients - Retrospective Double Center Study
Brief Title: Epidemiology of Bacteremia at Two Tertiary ICUs in Switzerland
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02302
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia | interventions — Blood Culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bern ICU
  Interventions: Diagnostic Test: Blood Culture
- Lausanne ICU
  Interventions: Diagnostic Test: Blood Culture

INTERVENTIONS:
Diagnostic Test: Blood Culture — Blood Culture

SUMMARY:
The objectives of the retrospective cohort study is to describe the actual current practice of antibiotic treatment duration for bloodstream infections in critically ill patients at two tertiary hospitals (ICU Inselspital Bern and ICU CHUV Lausanne), to examine patient, pathogen and infectious syndrome factors associated with selection of shortened treatment duration, and to describe the expected time course of clinical resolution among bacteremic patients.

ELIGIBILITY:
Inclusion Criteria:

Patient has a positive blood culture with a pathogenic organism Patient is critically ill at the time the blood culture was collected as defined by the following:

1. was treated at the ICU/IMC at the time of blood culture collection;
2. or has been admitted to ICU/IMC in the 48 hours after blood culture collection

Exclusion Criteria:

1. Patient has a single positive blood culture with a common contaminant organism:

   * coagulase negative staphylococci;
   * Bacillus spp.;
   * Corynebacterium spp.;
   * Propionibacterium spp.;
   * Aerococcus spp.;
   * Micrococcus spp.
2. Explicit documentation that the patient does not want to participate in any study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient is critically ill at the time the blood culture was collected and was treated at the ICU/IMC at the time of blood culture collection or has been admitted to ICU/IMC in the 48 hours after blood culture collection.
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Antibiotic Treatment Duration | Hospital discharge, expected to be on average ca. 15-20 days
  Days of adequate antibiotic treatment in Patients with Bacteremia

SECONDARY OUTCOMES:
Days of ICU stay | ICU discharge, expected to be on average ca. 5-15 days
  Days of ICU Stay in Patients with Bacteremia
Days of hospital stay | Hospital discharge, expected to be on average ca. 15-25 days
  Days of Inhospital Stay in Patients with Bacteremia

CONTACTS AND LOCATIONS:
Overall Officials: Josef Prazak, MD, PhD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Departement of Intensive Care Medicine, Bern, Switzerland

REFERENCES:
- [Derived] Zuercher P, Moser A, Frey MC, Pagani JL, Buetti N, Eggimann P, Daneman N, Fowler R, Que YA, Prazak J. The effect of duration of antimicrobial treatment for bacteremia in critically ill patients on in-hospital mortality - Retrospective double center analysis. J Crit Care. 2023 Apr;74:154257. doi: 10.1016/j.jcrc.2023.154257. Epub 2023 Jan 23. PMID 36696827